CLINICAL TRIAL: NCT00254722
Title: Safety of Autologous Stem Cell Treatment for Traumatic Brain Injury in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Charles Cox, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-05-0004; 1R21HD042659-01A1 (NIH)
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Stem Cell
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): single arm study
  Interventions: Drug: Autologous bone marrow precursor cell harvest and transplant

INTERVENTIONS:
Drug: Autologous bone marrow precursor cell harvest and transplant — Bone marrow harvest (3 ml/kg of body weight) performed between 12 and 30 hours post injury, followed by single intravenous infusion of bone marrow progenitor cells - target dose is 6x10^6 mononuclear cells/kg body weight, administered within 36 hours of injury

SUMMARY:
The purpose of this study is to determine if bone marrow progenitor cell (BMPC) autologous transplantation in children after isolated traumatic brain injury is safe and will improve functional outcome.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) contributes to 50% of all trauma deaths. The mortality rate for children following severe TBI (Glasgow Coma Scale < 9) ranges from 14-24%. There is currently no therapy to reverse the primary injury associated with TBI. Bone marrow precursor cells (BMPC) or bone marrow mononuclear cellular fractions of bone marrow contain mesenchymal stem cells (MSC) and hematopoetic stem cells (HSC). These cells are a component of bone marrow that preferentially migrate to the site of brain injury and differentiate into neurons and cell supporting elements, improving functional outcome in animals. The primary objective of this study is to determine if BMPC harvest and autologous transplantation is safe in children after TBI. The secondary objective is to determine if late functional outcome is improved with BMPC autologous transplantation compared to age and severity matched concomitant controls. Safety will be determined by monitoring cerebral and systemic hemodynamics during harvest and transplantation, neurologic events (seizure, change in GCS, stroke), local site inflammation/injury, and secondary organ injury. Late outcomes will be determined using age-corrected Glasgow Outcome Scores, and a battery of functional outcome measures. In vitro, an aliquot of cells harvested from patients will be studied for labeling with magnetodendrimers as a feasibility study, and these cells will not be reinfused into the patients. The primary endpoint is to assess the safety of autologous BMPC harvest/transplantation in the acute injury phase (hospital stay) and the secondary endpoint is to assess efficacy through 1 and 6 month post-injury follow-up. The rationale for the use of autologous BMPC transplantation is based on a large volume of in vitro and in vivo animal data (see background and significance section). The rationale for using children as the primary population is that children have a greater neurologic plasticity with a unique injury pattern when compared to adults. Children are more likely to have isolated TBI that is more diffuse and less likely to be secondary to extra-axial fluid collections. Patients aged 5-14 years old with GCS of 5-8 will be considered for enrollment into the study. Within 24-36 hours of injury, enrolled patients will undergo bone marrow harvest/BMPC separation and re-infusion. Daily monitoring of the safety outcomes measures and long term neurologic outcomes will be performed. This study should determine if bone marrow harvest, BMPC separation, and reinfusion is safe in children after severe TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Between 5 and 14 years of age on the day of injury
2. Hospital admission Glasgow coma score between 5 and 8
3. Initial injury occurring less than 24 hours prior to consent

Exclusion Criteria:

1. Known history of:

   * Previous brain injury
   * Developmental delay
   * Neurologic impairment and/or deficit
   * Seizure disorder requiring anti-convulsant therapy
   * Renal disease or altered renal function as defined by serum creatinine > 1.5 mg/dL at admission
   * Hepatic disease or altered liver function as defined by SGPT > 150 U/L, and/or T. bilirubin > 1.3 mg/dL at admission
   * Cancer
   * Immunosuppression as defined by WBC < 3 (10x3) at admission
   * HIV
2. Obliteration of perimesencephalic cistern on initial head CT/MRI suggesting prolonged hypoxic ischemic insult
3. Initial hospital ICP > 40
4. Hemodynamic instability at the time of consent defined as ongoing fluid resuscitation and/or requirement for inotropic support to maintain MAP at or above normals for age - does not include CPP based inotropic support
5. Uncorrected coagulopathy at the time of consent defined as INR > 1.4; PTT > 35 sec; PLT < 100,000; fibrinogen < 100 g/dL
6. Unstable pelvic fractures defined as requiring operative fixation to manage
7. Pulmonary contusions defined as a chest x-ray with non-anatomic opacification and/or PaO2:FIO2 ratio < 250 associated with the mechanism or injury
8. Solid or hollow visceral injury of the abdomen and/or pelvis as diagnosed by CT or other imaging
9. Spinal cord injury as diagnosed by CT or MR imaging or by clinical findings.
10. Persistent hypoxia defined as SaO2 < 94% for > 30 minutes occurring at any time from hospital admission to time of consent
11. Positive urine pregnancy test
12. Participation in an intervention study
13. Unwillingness to return for follow-up visits

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2006-04; Primary Completion 2008-11 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
neurologic events [seizures, change in Glasgow coma scale (GCS), cerebral vascular accident (CVA)] | 12 hours post cellular product infusion, up to 21 days post infusion
infectious morbidity | up to 21 days post cellular product infusion
secondary organ injury | up to 21 days post cellular product infusion

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Cox, Jr., M.D., Principal Investigator — The University of Texas Health Science Center, Houston